CLINICAL TRIAL: NCT04643808
Title: Noninvasive Brain Stimulation to Improve Oromotor Function In Neonates With Advanced Neuroimaging to Determine Safety and Target Engagement of taVNS for Neurorehabilitation
Brief Title: taVNS Paired With Bottle Feeding in Infants Failing Oral Feeds
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dorothea D. Jenkins, Professor of Pediatrics, Medical University of South Carolina
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 67997; P20GM109040 (NIH); P2CHD086844 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-11-25 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Poor Feeding; Infant Development; Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study investigators delivered taVNS once or twice a day during a bottle feed for 2 weeks. Stimulation was paired with nutritive sucking and swallowing, and was paused during rest or burping. If PO feeds had not progressed after 2 weeks of taVNS treatment, the parents and the clinical team made decisions about timing of G-tube placement. If substantial progress in po feeds was made during the treatment period, but the infant was not quite to full oral feeds, the clinical team and parents could elect to continue for 1-2 weeks.
Who Masked: Outcomes Assessor
Masking Description: Co-investigators analyzing diffusion MRI data were blinded to the timing of the MRI scans (pre- and post-treatment) and dose of taVNS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- taVNS once daily (Experimental): taVNS paired with bottle feeding once daily for 2-3 weeks
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- taVNS twice daily (Experimental): taVNS paired with bottle feeding twice daily for 2-3 weeks
  Interventions: Device: transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Microcurrent stimulation delivered to the left tragus, with stimulation 'on' during sucking from a bottle, and 'off' at rest during bottle feeding
  Other Names: taVNS

SUMMARY:
Oromotor dysfunction and poor feeding is common after premature birth and hypoxic ischemic encephalopathy (HIE). Pairing vagus nerve stimulation (VNS) with motor activity accelerates functional improvements after stroke. This study is designed to investigate whether transcutaneous auricular VNS (taVNS) paired with oromotor rehabilitation is tolerable, safe, and facilitates motor learning in infants who have failed oral feeding.

DETAILED DESCRIPTION:
Feeding difficulty is the primary reason for delayed hospital discharge from the neonatal intensive care unit (NICU), with increased hospital costs and a negative impact on neurodevelopment. Occupational or speech therapists typically start oral stimulation programs early, then feed infants by mouth (PO) daily to encourage safe feeding while learning this motor skill. Even after weeks or months of rehabilitation with therapists, many infants need a gastrostomy tube (G-tube) surgically placed for adequate nutrition. With improved survival rates of more critically ill neonates, the national rate of G-tube placement has doubled from 2000-2012.

Difficulty learning the motor sequence for oral feeding may be due to brain injury from infection, ischemia, and dysmaturity. In these infants, the normal integrative connectivity that occurs after birth between the cortex, basal ganglia, and brainstem may be disturbed, resulting in poor coordination and failure to learn the complex motor task of feeding, when it should be a normal reflex. Therapies that facilitate motor learning and enhance feeding skills would have a significant impact for infants who fail feeding rehabilitation.

In neonates with brain dysmaturity or overt brain injury, neuromodulation of abnormal circuits may positively boost neuronal connectivity and enhance neuroplasticity. Vagus nerve stimulation (VNS) paired with motor activity facilitates cortical reorganization and neurogenesis, and improves motor function in animal stroke models. A noninvasive form of VNS, transcutaneous auricular VNS (taVNS), targets the auricular branch of the vagus nerve to activate vagal afferent and efferent networks. In adult patients with limb impairment after brain injury, pairing taVNS with motor activation is safe, enhances plasticity and improves functional motor recovery. This work in adult humans extends and supports the animal evidence that pairing VNS with a motor or behavioral intervention restores brain function.

The study investigators applied the model of taVNS paired with a motor behavior to infants in the NICU in a prospective, open-label trial exploring the use of once and twice daily taVNS-paired rehabilitation training to enhance oral feeding in infants who are failing oral feeds and slated to receive a G-tube.

After obtaining informed consent, MRIs are obtained before starting treatment, and at end of 2-3 week treatment period. In a subset of 10 patients the study investigators also obtain modified barium swallows prior to and after the treatment period, with taVNS on and off during swallowing. Daily feeding volumes as well as the slope of change of po feeding volumes are recorded before and after starting taVNS.

ELIGIBILITY:
Inclusion Criteria:

* Infants must be clinically stable, on minimal respiratory support (nasal cannula, or room air), are not restricted for attempting every feed by mouth, and are currently failing oral feeding such that the clinical team is broaching gastrostomy tube (G-tube) placement with the parents. The infant will be greater than or equal to 39weeks gestation at enrollment and either

  1. Premature at birth and attempting oral feeds for at least 3 weeks or
  2. Infants who are neart-term or term at birth, with significant medical issues that have precluded oral feeding, such as hypoxic ischemic encephalopathy (HIE), and attempting oral feeds for at least 2 weeks.

Exclusion Criteria:

* Unstable infants or those requiring positive pressure respiratory support.
* Infants <38weeks gestation at enrollment.
* Major unrepaired congenital anomalies or anomalies that limit feeding volumes
* Cardiomyopathy
* Repeated episodes of autonomic instability (apnea or bradycardia) which are not self resolving

Ages: 3 Weeks to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Jenkins, MD, Principal Investigator — Medical University of South Carolina; Bashar Badran, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Badran BW, Jenkins DD, DeVries WH, Dancy M, Summers PM, Mappin GM, Bernstein H, Bikson M, Coker-Bolt P, George MS. Transcutaneous auricular vagus nerve stimulation (taVNS) for improving oromotor function in newborns. Brain Stimul. 2018 Sep-Oct;11(5):1198-1200. doi: 10.1016/j.brs.2018.06.009. Epub 2018 Jun 30. No abstract available. PMID 30146041
- [Result] Badran BW, Jenkins DD, Cook D, Thompson S, Dancy M, DeVries WH, Mappin G, Summers P, Bikson M, George MS. Transcutaneous Auricular Vagus Nerve Stimulation-Paired Rehabilitation for Oromotor Feeding Problems in Newborns: An Open-Label Pilot Study. Front Hum Neurosci. 2020 Mar 18;14:77. doi: 10.3389/fnhum.2020.00077. eCollection 2020. PMID 32256328
- [Result] Cook DN, Thompson S, Stomberg-Firestein S, Bikson M, George MS, Jenkins DD, Badran BW. Design and validation of a closed-loop, motor-activated auricular vagus nerve stimulation (MAAVNS) system for neurorehabilitation. Brain Stimul. 2020 May-Jun;13(3):800-803. doi: 10.1016/j.brs.2020.02.028. Epub 2020 Feb 27. PMID 32289710
- [Derived] Jenkins DD, Moss HG, Adams LE, Hunt S, Dancy M, Huffman SM, Cook D, Jensen JH, Summers P, Thompson S, George MS, Badran BW. Higher Dose Noninvasive Transcutaneous Auricular Vagus Nerve Stimulation Increases Feeding Volumes and White Matter Microstructural Complexity in Open-Label Study of Infants Slated for Gastrostomy Tube. J Pediatr. 2023 Nov;262:113563. doi: 10.1016/j.jpeds.2023.113563. Epub 2023 Jun 16. PMID 37329979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neonatal intensive Care Unit
Period: Overall Study
Arm/Group | taVNS Once Daily | taVNS Twice Daily
Started | 14 | 21
Completed | 14 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- taVNS Once Daily: taVNS paired with bottle feeding once daily for 2-3 weeks
  Infants born preterm or near term/term HIE infants who failed to make progress in PO volumes, and were clinically determined to require a G-tube due to failure to achieve oral feeds sufficient for discharge from the hospital.
- taVNS Twice Daily: taVNS paired with bottle feeding twice daily for 2-3 weeks
  Infants born preterm or near term/term HIE infants who failed to make progress in PO volumes, and were clinically determined to require a G-tube due to failure to achieve oral feeds sufficient for discharge from the hospital.
- Total: Total of all reporting groups
Arm/Group | taVNS Once Daily | taVNS Twice Daily | Total
Number analyzed (Participants) | 14 | 21 | 35
Age, Continuous [Mean (Standard Deviation); unit: post menstrual age in months ofgestation] — post menstrual age in weeks gestation at enrollment
  post menstrual age in months ofgestation | 44 (4.8) | 42.1 (2.8) | 42.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 20 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
change in ml/kg/d po [Mean (Standard Deviation); unit: ml/kg/d consumed orally (po)] — Population: averaged over 7days prior to starting taVNS treatment
  ml/kg/d consumed orally (po) | -0.6 (4.8) | 0.03 (3.6) | -0.23 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants Who Took All Feeds by Mouth (Responders)
Description: Number of infants who maintained full daily PO intake for 4 days (>120 ml/kg/day) and gained weight adequate for discharge (>20 g/day) were classified as 'Responders'.
Time Frame: 3 weeks
Population: Responders who achieved full oral feeds and weight gain adequate for discharge
Measure: Count of Participants; unit: Participants
Arm/Group | taVNS Once Daily | taVNS Twice Daily
Number analyzed (Participants) | 14 | 21
Participants | 8 | 11

2. Primary Outcome: ml/kg/d Increase Over 7d During taVNS
Description: The change in ml/kg/d of oral feeds over the 7 days during taVNS-paired feeds
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ml/kg/d increase over 7d
Arm/Group | taVNS Once Daily | taVNS Twice Daily
Number analyzed (Participants) | 14 | 21
ml/kg/d increase over 7d | 3.9 (4.2) | 6.0 (4.16)

3. Primary Outcome: Neuroplasticity as Measured by the Change in White Matter Tract Integrity Via Fractional Anisotropy
Description: changes in radial kurtosis diffusion in Corticospinal tracts at the cerebellar peduncles assessed per week of treatment, change from baseline to week 3 reported. Kurtosis is a dimensionless summary statistic that quantifies the amount of non-Gaussianity within the tissue on a scale from 0 to infinity. Higher values indicate greater complexity in the white matter tract. The scale has no title other than diffusion kurtosis.
Time Frame: change from baseline to week 3
Measure: Mean (Standard Deviation); unit: kurtosis units on a scale
Groups:
- taVNS Responders: all taVNS (1X+2X) who attained full oral feeds
- taVNS Non-responders: all taVNS (1X+2X) who did not attain full oral feeds and required a Gtube for feeds
Arm/Group | taVNS Responders | taVNS Non-responders
Number analyzed (Participants) | 9 | 11
kurtosis units on a scale | 0.07 (.02) | 0.02 (.02)

4. Secondary Outcome: Number of Episodes of Bradycardia
Description: bradycardic episodes = heart rate <80 beats per minute for 5 seconds
Time Frame: 3 weeks, during taVNS sessions
Measure: Number; unit: bradycardic events
Arm/Group | taVNS Once Daily | taVNS Twice Daily
Number analyzed (Participants) | 14 | 21
bradycardic events | 1 | 0

5. Secondary Outcome: Number of Treatment Sessions With Sustained Increase in 'Neonatal and Infant Pain Scale' (NIPS) Scores During taVNS
Description: Number of treatment sessions with sustained increase of 3 points in Neonatal and Infant Pain Scale (NIPS) scores from before to during taVNS: NIPS recorded at before, midway, and at the end of each treatment session. NIPS scores range from 0 (no discomfort) to 7 (maximum discomfort). An increase of 3 points on the NIPS scale indicates more discomfort with stimulation.
Time Frame: 30min treatment session
Population: total number of treatment sessions for all participants
Measure: Count of Units; unit: treatment sessions
Units Other Than Participants: treatment sessions
Arm/Group | taVNS Once Daily | taVNS Twice Daily
Number analyzed (Participants) | 14 | 21
Number analyzed (treatment sessions) | 228 | 623
treatment sessions | 3 | 0

ADVERSE EVENTS:
Time Frame: over the 2-3 weeks of the taVNS-paired feeds
Description: we monitored every session for adverse events and for SAE of receiving Gtube or death after discharge
Arm/Group | taVNS Once Daily | taVNS Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/14 | 0/21

LIMITATIONS AND CAVEATS:
no concurrent control group, open label dose study (not randomized)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04643808/Prot_SAP_000.pdf